CLINICAL TRIAL: NCT04047563
Title: A Prospective, Multicentric, Randomized, Double-blind, Parallel, Phase III Clinical Study to Assess Efficacy of PMZ-1620 Along With Standard Treatment in Patients of Acute Ischemic Stroke
Brief Title: Efficacy of Sovateltide (PMZ-1620) in Patients of Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-1620/CT-3.1/2019
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Ischemia; Cerebral Infarction; Stroke, Acute
Keywords: Endothelin; Neurogenesis; Neural progenitor cells
MeSH Terms: conditions — Brain Ischemia; Cerebral Infarction; Stroke | interventions — sovateltide

STUDY DESIGN:
Intervention Model Description: In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1, 3, and day 6 (total dose/day: 0.9 µg/kg body weight).
  In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, 3 and day 6 post randomization.
  In both treatment groups, subjects will be provided the best available standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline + Standard of care (Active Comparator): Patients will receive the best available standard of care. In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, 3 and day 6 post randomization.
  Interventions: Drug: Normal Saline along with standard treatment
- PMZ-1620 (sovateltide) + Standard of care (Experimental): Patients will receive the best available standard of care. In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1, 3, and day 6 (total dose/day: 0.9 µg/kg body weight).
  Interventions: Drug: PMZ-1620 (sovateltide) along with standard treatment

INTERVENTIONS:
Drug: Normal Saline along with standard treatment — PMZ-1620 (sovateltide) is an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in cerebral ischemic stroke patients. In this arm normal saline along with standard treatment will be given for active comparison.
  Other Names: Vehicle
  Arms: Normal Saline + Standard of care
Drug: PMZ-1620 (sovateltide) along with standard treatment — PMZ-1620 (sovateltide) is an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in cerebral ischemic stroke patients.
  Other Names: PMZ-1620
  Arms: PMZ-1620 (sovateltide) + Standard of care

SUMMARY:
In the present prospective, multicentric, randomized, double-blind, parallel, saline-controlled phase II clinical study; the investigators plan to evaluate the efficacy of sovateltide (IRL-1620 or PMZ-1620) therapy along with standard supportive care in patients of acute ischemic stroke.

DETAILED DESCRIPTION:
The peptide Sovateltide (IRL-1620) is a highly selective ETB receptor agonist. There are hidden stem cells in the brain, which becomes active following injury to the brain. Intravenous administration of PMZ-1620 (sovateltide) augments the activity of neuronal progenitor cells in the brain to repair the damage by formation of new mature neurons and blood vessels. In addition, PMZ-1620 has anti-apoptotic activity and also increases cerebral blood flow when administered following ischemia. It was discovered that in rat model of ischemic stroke, sovateltide, significantly improved survival, reduces neurological and motor function deficit while effectively decreasing infarct volume, edema and oxidative stress. The convincing results of preclinical efficacy studies of Sovateltide in ischemic stroke and its safety affirmation from phase I and phase II clinical studies encouraged us to investigate its efficacy in human patients of ischemic stroke. In the present prospective, multicentric, randomized, double-blind, parallel, saline-controlled phase II clinical study; the investigators plan to evaluate the efficacy of Sovateltide therapy along with standard supportive care in patients of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females Aged 18 years through 78 years (have not had their 79th birthday).
2. Patient or Legally Authorized Representative willing to give informed Consent before study procedure.
3. Stroke is ischemic in origin and radiologically confirmed Computed Tomography (CT) scan or diagnostic magnetic resonance imaging (MRI) prior to enrolment. No hemorrhage as proved by cerebral CT/MRI scan.
4. Cerebral ischemic stroke patients presenting upto 24 hours after onset of symptoms with mRS score of 3-4 (pre-stroke mRS score of 0 or 1) and NIHSS score >5 (NIHSS Level of Consciousness (1A) score must be < 2). This also includes patients who had ischemic stroke in the past and are completely recovered from earlier episode before having new or fresh stroke.
5. Patient is < 24 hours from time of stroke onset when the first dose of PMZ-1620 therapy is administered. Time of onset is when symptoms began; for stroke that occurred during sleep, time of onset is when patient was last seen or was self- reported to be normal.
6. Reasonable expectation of availability to receive the full PMZ-1620 course of therapy, and to be available for subsequent follow-up visits.

Exclusion Criteria:

1. Patients receiving endovascular therapy or is a candidate for any surgical intervention for treatment of stroke which may include but not limited to endovascular techniques.
2. Patients classified as comatose, defined as a patient who required repeated stimulation to attend, or is obtunded and requires strong or painful stimulation to make movements (NIHSS Level of Consciousness (1A) score ≥ 2).
3. Evidence of intracranial hemorrhage (intracerebral hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hemorrhage, acute or chronic subdural hematoma on the baseline CT or MRI scan.
4. Known pregnancy.
5. Confounding pre-existing neurological or psychiatric disease.
6. Concurrent participation in any other therapeutic clinical trial.
7. Evidence of any other major life-threatening or serious medical condition that would prevent completion of the study protocol, impair the assessment of outcome, or in which PMZ-1620 therapy would be contraindicated or might cause harm to the patient.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Change in National Institute of Health Stroke Scale (NIHSS) | 90 days
  Neurological outcome as assessed by National Institute of Health Stroke Scale (NIHSS) score post randomization. NIHSS is 42 point scale where 0 is the best and 42 is the worst outcome.
Change in modified Rankin Scale (mRS) | 90 days
  Neurological outcome as assessed by modified Rankin Scale (mRS) score post randomization. mRS is a 7 grade scale from 0 to 6, where 0 is the best and 6 is the worst outcome.
Change in Barthel index [BI] | 90 days
  Overall clinical outcome as assessed by Barthel index [BI] scores) at 3 months post randomization. BI is a 10 item scale with scores ranging from 0 to 100, where a score of 100 is the best and 0 is the worst outcome.
Change in the proportion of ischemic stroke patients with NIHSS score <6 | 90 days
  Change in the proportion of ischemic stroke patients with National Institute of Health Stroke Scale (NIHSS) score <6 at day 6, 1 month and 3 months. NIHSS is 42 point scale where 0 is the best and 42 is the worst outcome.
Change in the proportion of ischemic stroke patients with mRS score <2 | 90 days
  Change in the proportion of ischemic stroke patients with modified Rankin Scale (mRS) score <2 at day 6, 1 month and 3 months. mRS is a 7 grade scale from 0 to 6, where 0 is the best and 6 is the worst outcome.
Change in the proportion of ischemic stroke patients with Barthel index (BI) score >60 | 90 days
  Change in the proportion of ischemic stroke patients with Barthel index (BI) score >60 at day 6, 1 month and 3 months. BI is a 10 item scale with scores ranging from 0 to 100, where a score of 100 is the best and 0 is the worst outcome.

SECONDARY OUTCOMES:
Change in Quality-of-life as assessed by EuroQol-EQ-5D | 90 days
  Quality-of-life as assessed by EuroQol-EQ-5D will be determined at 1 month and 3 months post randomization. EuroQol-EQ-5D is a concise, generic instrument that could be used to measure, compare and value health status across disease areas. It is a five dimension instrument with scores ranging from 0 to 100, where a score of 100 is the best and 0 is the worst outcome.
Change in Stroke-Specific Quality of Life (SSQOL) | 90 days
  Stroke-Specific Quality of Life (SSQOL) will be assessed at 1 month and 3 months post randomization. SSQOL is composed of 49 items with scores ranging from 49 to 245, where a score of 245 is the best and 49 is the worst outcome.
Incidence in recurrence of ischemic stroke | 90 days
  Incidence of recurrent ischemic stroke within 1 month and 3 months post-randomization, as assessed by Questionnaire to Validate Stroke-Free Status
Incidence of mortality | 90 days
  Incidence of mortality within 3 months post-randomization
Incidence of Intra-Cerebral Hemorrhage (ICH) | 30 hours
  Incidence of symptomatic Intra Cerebral Hemorrhage (ICH) within 24 (± 6) hours of randomization
Incidence of PMZ-1620 related adverse events | 90 days
  Another objective of the study is to determine incidence of drug (PMZ-1620) related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, MD, PhD, Study Chair — Chairman and CEO
Locations (11):
- India (11):
  - Pushpanjali Hospital & Research Centre Pvt. Ltd, Agra, Uttar Pradesh
  - Radiant Superspeciality Hospital, Amravati
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Lalitha Superspecialities Hospital, Guntur
  - Dayanand Medical College & Hospital, Ludhiana
  - Department of Neurology, Christian Medical College and Hospital, Ludhiana
  - Sidhu Hospital Pvt. Ltd., Ludhiana
  - New Era Hospital & Research Institute, Nagpur
  - Chopda Medicare & Research Centre, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Indian Spinal Injury Centre, New Delhi

IPD SHARING:
Plan to Share IPD: No
Results will be communicated and published as manuscript

REFERENCES:
- [Background] Briyal S, Ranjan AK, Hornick MG, Puppala AK, Luu T, Gulati A. Anti-apoptotic activity of ETB receptor agonist, IRL-1620, protects neural cells in rats with cerebral ischemia. Sci Rep. 2019 Jul 18;9(1):10439. doi: 10.1038/s41598-019-46203-x. PMID 31320660
- [Background] Cifuentes EG, Hornick MG, Havalad S, Donovan RL, Gulati A. Neuroprotective Effect of IRL-1620, an Endothelin B Receptor Agonist, on a Pediatric Rat Model of Middle Cerebral Artery Occlusion. Front Pediatr. 2018 Oct 23;6:310. doi: 10.3389/fped.2018.00310. eCollection 2018. PMID 30406063
- [Background] Gulati A, Hornick MG, Briyal S, Lavhale MS. A novel neuroregenerative approach using ET(B) receptor agonist, IRL-1620, to treat CNS disorders. Physiol Res. 2018 Jun 27;67(Suppl 1):S95-S113. doi: 10.33549/physiolres.933859. PMID 29947531
- [Background] Bhalla S, Leonard MG, Briyal S, Gulati A. Distinct Alteration in Brain Endothelin A and B Receptor Characteristics Following Focal Cerebral Ischemia in Rats. Drug Res (Stuttg). 2016 Apr;66(4):189-95. doi: 10.1055/s-0035-1559779. Epub 2015 Sep 23. PMID 26398673
- [Background] Leonard MG, Gulati A. Endothelin B receptor agonist, IRL-1620, enhances angiogenesis and neurogenesis following cerebral ischemia in rats. Brain Res. 2013 Aug 28;1528:28-41. doi: 10.1016/j.brainres.2013.07.002. Epub 2013 Jul 11. PMID 23850649
- [Background] Leonard MG, Briyal S, Gulati A. Endothelin B receptor agonist, IRL-1620, provides long-term neuroprotection in cerebral ischemia in rats. Brain Res. 2012 Jun 29;1464:14-23. doi: 10.1016/j.brainres.2012.05.005. Epub 2012 May 9. PMID 22580085
- [Background] Leonard MG, Briyal S, Gulati A. Endothelin B receptor agonist, IRL-1620, reduces neurological damage following permanent middle cerebral artery occlusion in rats. Brain Res. 2011 Oct 28;1420:48-58. doi: 10.1016/j.brainres.2011.08.075. Epub 2011 Sep 7. PMID 21959172
- [Background] Ranjan AK, Briyal S, Gulati A. Sovateltide (IRL-1620) activates neuronal differentiation and prevents mitochondrial dysfunction in adult mammalian brains following stroke. Sci Rep. 2020 Jul 29;10(1):12737. doi: 10.1038/s41598-020-69673-w. PMID 32728189
- [Background] Ranjan AK, Briyal S, Khandekar D, Gulati A. Sovateltide (IRL-1620) affects neuronal progenitors and prevents cerebral tissue damage after ischemic stroke. Can J Physiol Pharmacol. 2020 Sep;98(9):659-666. doi: 10.1139/cjpp-2020-0164. Epub 2020 Jun 23. PMID 32574518
- [Result] Gulati A, Agrawal N, Vibha D, Misra UK, Paul B, Jain D, Pandian J, Borgohain R. Safety and Efficacy of Sovateltide (IRL-1620) in a Multicenter Randomized Controlled Clinical Trial in Patients with Acute Cerebral Ischemic Stroke. CNS Drugs. 2021 Jan;35(1):85-104. doi: 10.1007/s40263-020-00783-9. Epub 2021 Jan 11. PMID 33428177
- [Derived] Gulati A, Adwani SG, Vijaya P, Agrawal NR, Ramakrishnan TCR, Rai HP, Jain D, Sundarachary NV, Pandian JD, Sardana V, Sharma M, Sidhu GK, Anand SS, Vibha D, Aralikatte S, Khurana D, Joshi D, Karadan U, Siddiqui MSI. Efficacy and Safety of Sovateltide in Patients with Acute Cerebral Ischaemic Stroke: A Randomised, Double-Blind, Placebo-Controlled, Multicentre, Phase III Clinical Trial. Drugs. 2024 Dec;84(12):1637-1650. doi: 10.1007/s40265-024-02121-5. Epub 2024 Nov 15. PMID 39542995